CLINICAL TRIAL: NCT00499733
Title: Sequential Administration of Cryoablation and Cyclophosphamide for Advanced Solid Epithelial Cancer
Brief Title: Cyclophosphamide and Cryoablation in Treating Patients With Advanced or Metastatic Epithelial Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study was terminated per PI decision.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0685; P30CA006973 (NIH); NA_00003073 (Other: JHM IRB); JHOC-J0685; CDR0000554417 (Other: other)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2017-02

CONDITIONS: Cancer
Keywords: carcinoma of unknown primary; recurrent carcinoma of unknown primary; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer; male breast cancer; recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; chondrosarcoma; metastatic osteosarcoma; recurrent osteosarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; previously treated childhood rhabdomyosarcoma; recurrent childhood rhabdomyosarcoma; metastatic childhood soft tissue sarcoma; recurrent childhood soft tissue sarcoma; ovarian sarcoma; stage IIIB uterine sarcoma; stage IIIC uterine sarcoma; stage IIIA uterine sarcoma; stage IVA uterine sarcoma; stage IVB uterine sarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; stage III colon cancer; stage IV colon cancer; recurrent colon cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; recurrent childhood liver cancer; stage III childhood liver cancer; stage IV childhood liver cancer; stage III pancreatic cancer; localized osteosarcoma; malignant giant cell tumor of bone; stage IV melanoma; recurrent melanoma; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage III basal cell carcinoma of the lip; stage III squamous cell carcinoma of the lip and oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; high-grade salivary gland mucoepidermoid carcinoma; salivary gland adenocarcinoma; salivary gland adenoid cystic carcinoma; salivary gland anaplastic carcinoma; salivary gland malignant mixed cell type tumor; salivary gland poorly differentiated carcinoma; salivary gland squamous cell carcinoma; low-grade salivary gland mucoepidermoid carcinoma; salivary gland acinic cell tumor; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent salivary gland cancer; intraocular lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent pancreatic cancer; recurrent uterine sarcoma; newly diagnosed carcinoma of unknown primary; advanced adult primary liver cancer; ciliary body and choroid melanoma, medium/large size; conjunctival melanoma; stage IV pancreatic cancer; stage IIIA melanoma; stage IIIB melanoma; stage IIIC melanoma; tongue cancer; stage IIIA intraocular melanoma; stage IIIB intraocular melanoma; stage IIIC intraocular melanoma; stage IV intraocular melanoma
MeSH Terms: conditions — Neoplasms; Neoplasms, Unknown Primary; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Renal Cell; Prostatic Neoplasms; Breast Neoplasms, Male; Breast Neoplasms; Chondrosarcoma; Osteosarcoma; Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Colonic Neoplasms; Carcinoma, Hepatocellular; Pancreatic Neoplasms; Melanoma; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms; Intraocular Lymphoma; Uveal Melanoma; Tongue Neoplasms | interventions — Cyclophosphamide; Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Intervention (Experimental): Participant will receive one time intravenous infusion of cyclophosphamide three days after scheduled cryoablation surgery.
  Interventions: Drug: cyclophosphamide; Device: Cryoablation

INTERVENTIONS:
Drug: cyclophosphamide — 500 mg/m^2 of cyclophosphamide is infused via intravenous route three days post cryoablation surgery.
  Other Names: cytoxan
Device: Cryoablation — Per treating physician's discretion, largest and most accessible lesion will be treated with cryoablation surgery on day 0 of the study.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Cryoablation kills cancer cells by freezing them. Giving chemotherapy together with cryoablation may kill more cancer cells.

PURPOSE: This clinical trial is studying how well giving cyclophosphamide together with cryoablation works in treating patients with advanced or metastatic epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Document radiologic and/or tumor marker response to cryotherapy of tumor lesions followed by cyclophosphamide.

OUTLINE: This is a pilot study.

Patients undergo percutaneous biopsy of the targeted lesion prior to cryoablation. Patients then undergo percutaneous or open cryotherapy of the largest or most accessible lesion on day 0. On day 3, patients receive cyclophosphamide IV over 1 hour.

Tumor markers (if applicable) are assessed at baseline and monthly during study until marker progression.

After completion of study therapy, patients are followed periodically for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of epithelial solid tumors of any of the following sites or types:

  * Lung (closed to accrual as of 4/2/2009)
  * Renal
  * Prostate
  * Breast (closed to accrual as of 4/2/2009)
  * Sarcoma (closed to accrual as of 4/2/2009)
  * Colon (closed to accrual as of 4/2/2009)
  * Liver(closed to accrual as of 4/2/2009)
  * Pancreatic (closed to accrual as of 4/2/2009)
  * Bone (closed to accrual as of 4/2/2009)
  * Head and neck (closed to accrual as of 4/2/2009)
  * Melanoma (closed to accrual as of 4/2/2009)
  * Carcinoma of unknown primary (closed to accrual as of 4/2/2009)
* Advanced or metastatic disease
* Ineligible for or unwilling to undergo surgical resection
* Eligible for cryotherapy but not expected to be cured by cryotherapy alone

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Creatinine < 2.5 mg/dL
* Platelet count >75,000/mm³
* INR< 1.5
* No known HIV positivity
* No active, uncontrolled infection
* Not pregnant
* Negative pregnancy test
* Women of childbearing potential must practice adequate contraception
* No debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal treatment and follow-up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2010-07 (Actual); Study Completion 2013-01-09 (Actual)

PRIMARY OUTCOMES:
Safety, in terms of absences of severe adverse events (SAE) and unacceptable toxicity | Two years

SECONDARY OUTCOMES:
Tumor response, according to RECIST criteria | Two years
  tumor response will be measured according to RECIST (Response Evaluation Criteria In Solid Tumors) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Rodriguez, MD, PhD, Principal Investigator — Brady Urological Institute at Johns Hopkins Hospital
Locations (1):
- Brady Urological Institute at Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No